CLINICAL TRIAL: NCT03417050
Title: Synergy Between PCI With TAXUS and Cardiac Surgery: SYNTAX Extended Survival
Acronym: SYNTAXES
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Stuart Head, MD, PhD, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2016-716
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass grafting; percutaneous coronary intervention; drug eluting stent; survival status; long-term follow-up; complex coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Randomized CABG patients: Patients which were randomized to undergo CABG.
  Interventions: Other: No intervention will take place for this retrospective and observational study.
- Randomized PCI patients: Patients which were randomized to undergo PCI.
  Interventions: Other: No intervention will take place for this retrospective and observational study.
- Registry CABG: Patients for whom only one treatment option was suitable were included into a parallel, nested registry: the CABG registry for PCI-ineligible patients.
  Interventions: Other: No intervention will take place for this retrospective and observational study.
- Registry PCI: Patients for whom only one treatment option was suitable were included into a parallel, nested registry: the PCI registry for CABG-ineligible patients.
  Interventions: Other: No intervention will take place for this retrospective and observational study.

INTERVENTIONS:
Other: No intervention will take place for this retrospective and observational study. — No intervention will take place for this retrospective and observational study.

SUMMARY:
An investigator-driven, retrospective study to compare long-term survival-data (10-year follow-up) of patients with coronary artery disease (CAD), previously enrolled in the SYNTAX trial, who were randomized to percutaneous coronary intervention (PCI) using a paclitaxel (TAXUS) drug-eluting-stent (DES) or coronary artery bypass grafting (CABG).

ELIGIBILITY:
Patients which have previously been enrolled in the SYNTAX trial (randomized and registry patients)

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the SYNTAX trial and registries had to be diagnosed with three-vessel (3VD) or left main (LM) coronary artery disease. The vessels (diameter ≥1.5 mm and significant stenosis > 50%) deemed important to revascularize were determined by the Heart Team prior to randomization. The group of 3VD consists of patients with significant stenosis in vessels supplying all three major epicardial territories in absence of LM disease, as determined by the site investigators. The group of patients with LM disease consists of patients with a significant stenosis of the left main coronary artery, irrespective of additional vessel disease.
Sampling Method: Probability Sample
Enrollment: 2636 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Long-term survival status | 10-year
  All-cause death

SECONDARY OUTCOMES:
Cause of death | 10-year
  Cause-specific death, separated in cardiovascular and non-cardiovascular death with specific causes for cardiovascular deaths.

CONTACTS AND LOCATIONS:
Overall Officials: A. Pieter Kappetein, MD, PhD, Principal Investigator — Erasmus Medical Center; Friedrick W. Mohr, MD, PhD, Principal Investigator — German Heart Center, Leipzig, Germany; Patrick W.J.C. Serruys, MD, PhD, Principal Investigator — Imperial College London; Michael J. Mack, MD, PhD, Principal Investigator — Baylor Scott & White Health, Plano, TX, United States; David R. Holmes, MD, Principal Investigator — Mayo Clinic, Rochester, MN, United States; Marie-Claude Morice, MD, Principal Investigator — ICPS Ramsay-Generale de Sante, Massy, France; Piroze M. Davierwala, MD, Principal Investigator — German Heart Center, Leipzig, Germany; Stuart J. Head, MD, PhD, Principal Investigator — Erasmus Medical Center; Daniel J.F.M. Thuijs, MD, Study Chair — Erasmus Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sianos G, Morel MA, Kappetein AP, Morice MC, Colombo A, Dawkins K, van den Brand M, Van Dyck N, Russell ME, Mohr FW, Serruys PW. The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease. EuroIntervention. 2005 Aug;1(2):219-27. No abstract available. PMID 19758907
- [Background] Kappetein AP, Dawkins KD, Mohr FW, Morice MC, Mack MJ, Russell ME, Pomar J, Serruys PW. Current percutaneous coronary intervention and coronary artery bypass grafting practices for three-vessel and left main coronary artery disease. Insights from the SYNTAX run-in phase. Eur J Cardiothorac Surg. 2006 Apr;29(4):486-91. doi: 10.1016/j.ejcts.2006.01.047. Epub 2006 Feb 23. PMID 16497510
- [Background] Ong AT, Serruys PW, Mohr FW, Morice MC, Kappetein AP, Holmes DR Jr, Mack MJ, van den Brand M, Morel MA, van Es GA, Kleijne J, Koglin J, Russell ME. The SYNergy between percutaneous coronary intervention with TAXus and cardiac surgery (SYNTAX) study: design, rationale, and run-in phase. Am Heart J. 2006 Jun;151(6):1194-204. doi: 10.1016/j.ahj.2005.07.017. PMID 16781219
- [Background] Serruys PW, Morice MC, Kappetein AP, Colombo A, Holmes DR, Mack MJ, Stahle E, Feldman TE, van den Brand M, Bass EJ, Van Dyck N, Leadley K, Dawkins KD, Mohr FW; SYNTAX Investigators. Percutaneous coronary intervention versus coronary-artery bypass grafting for severe coronary artery disease. N Engl J Med. 2009 Mar 5;360(10):961-72. doi: 10.1056/NEJMoa0804626. Epub 2009 Feb 18. PMID 19228612
- [Background] Serruys PW, Onuma Y, Garg S, Sarno G, van den Brand M, Kappetein AP, Van Dyck N, Mack M, Holmes D, Feldman T, Morice MC, Colombo A, Bass E, Leadley K, Dawkins KD, van Es GA, Morel MA, Mohr FW. Assessment of the SYNTAX score in the Syntax study. EuroIntervention. 2009 May;5(1):50-6. doi: 10.4244/eijv5i1a9. PMID 19577983
- [Background] Banning AP, Westaby S, Morice MC, Kappetein AP, Mohr FW, Berti S, Glauber M, Kellett MA, Kramer RS, Leadley K, Dawkins KD, Serruys PW. Diabetic and nondiabetic patients with left main and/or 3-vessel coronary artery disease: comparison of outcomes with cardiac surgery and paclitaxel-eluting stents. J Am Coll Cardiol. 2010 Mar 16;55(11):1067-75. doi: 10.1016/j.jacc.2009.09.057. Epub 2010 Jan 14. PMID 20079596
- [Background] Girasis C, Serruys PW, Onuma Y, Colombo A, Holmes DR Jr, Feldman TE, Bass EJ, Leadley K, Dawkins KD, Morice MC. 3-Dimensional bifurcation angle analysis in patients with left main disease: a substudy of the SYNTAX trial (SYNergy Between Percutaneous Coronary Intervention with TAXus and Cardiac Surgery). JACC Cardiovasc Interv. 2010 Jan;3(1):41-8. doi: 10.1016/j.jcin.2009.10.019. PMID 20129567
- [Background] Garg S, Girasis C, Sarno G, Goedhart D, Morel MA, Garcia-Garcia HM, Bressers M, van Es GA, Serruys PW; SYNTAX trial investigators. The SYNTAX score revisited: a reassessment of the SYNTAX score reproducibility. Catheter Cardiovasc Interv. 2010 May 1;75(6):946-52. doi: 10.1002/ccd.22372. PMID 20146321
- [Background] Morice MC, Serruys PW, Kappetein AP, Feldman TE, Stahle E, Colombo A, Mack MJ, Holmes DR, Torracca L, van Es GA, Leadley K, Dawkins KD, Mohr F. Outcomes in patients with de novo left main disease treated with either percutaneous coronary intervention using paclitaxel-eluting stents or coronary artery bypass graft treatment in the Synergy Between Percutaneous Coronary Intervention with TAXUS and Cardiac Surgery (SYNTAX) trial. Circulation. 2010 Jun 22;121(24):2645-53. doi: 10.1161/CIRCULATIONAHA.109.899211. Epub 2010 Jun 7. PMID 20530001
- [Background] Mohr FW, Rastan AJ, Serruys PW, Kappetein AP, Holmes DR, Pomar JL, Westaby S, Leadley K, Dawkins KD, Mack MJ. Complex coronary anatomy in coronary artery bypass graft surgery: impact of complex coronary anatomy in modern bypass surgery? Lessons learned from the SYNTAX trial after two years. J Thorac Cardiovasc Surg. 2011 Jan;141(1):130-40. doi: 10.1016/j.jtcvs.2010.07.094. PMID 21168023
- [Background] Cohen DJ, Lavelle TA, Van Hout B, Li H, Lei Y, Robertus K, Pinto D, Magnuson EA, Mcgarry TF, Lucas SK, Horwitz PA, Henry CA, Serruys PW, Mohr FW, Kappetein AP. Economic outcomes of percutaneous coronary intervention with drug-eluting stents versus bypass surgery for patients with left main or three-vessel coronary artery disease: one-year results from the SYNTAX trial. Catheter Cardiovasc Interv. 2012 Feb 1;79(2):198-209. doi: 10.1002/ccd.23147. Epub 2011 Sep 26. PMID 21542113
- [Background] Kappetein AP, Feldman TE, Mack MJ, Morice MC, Holmes DR, Stahle E, Dawkins KD, Mohr FW, Serruys PW, Colombo A. Comparison of coronary bypass surgery with drug-eluting stenting for the treatment of left main and/or three-vessel disease: 3-year follow-up of the SYNTAX trial. Eur Heart J. 2011 Sep;32(17):2125-34. doi: 10.1093/eurheartj/ehr213. Epub 2011 Jun 22. PMID 21697170
- [Background] Morice MC, Feldman TE, Mack MJ, Stahle E, Holmes DR, Colombo A, Morel MA, van den Brand M, Serruys PW, Mohr F, Carrie D, Fournial G, James S, Leadley K, Dawkins KD, Kappetein AP. Angiographic outcomes following stenting or coronary artery bypass surgery of the left main coronary artery: fifteen-month outcomes from the synergy between PCI with TAXUS express and cardiac surgery left main angiographic substudy (SYNTAX-LE MANS). EuroIntervention. 2011 Oct 30;7(6):670-9. doi: 10.4244/EIJV7I6A109. PMID 21959312
- [Background] Mack MJ, Banning AP, Serruys PW, Morice MC, Taeymans Y, Van Nooten G, Possati G, Crea F, Hood KL, Leadley K, Dawkins KD, Kappetein AP. Bypass versus drug-eluting stents at three years in SYNTAX patients with diabetes mellitus or metabolic syndrome. Ann Thorac Surg. 2011 Dec;92(6):2140-6. doi: 10.1016/j.athoracsur.2011.06.028. Epub 2011 Oct 2. PMID 21967819
- [Background] Head SJ, Mack MJ, Holmes DR Jr, Mohr FW, Morice MC, Serruys PW, Kappetein AP. Incidence, predictors and outcomes of incomplete revascularization after percutaneous coronary intervention and coronary artery bypass grafting: a subgroup analysis of 3-year SYNTAX data. Eur J Cardiothorac Surg. 2012 Mar;41(3):535-41. doi: 10.1093/ejcts/ezr105. Epub 2011 Dec 21. PMID 22219412
- [Background] Arnold SV, Magnuson EA, Wang K, Serruys PW, Kappetein AP, Mohr FW, Cohen DJ; SYNTAX Investigators. Do differences in repeat revascularization explain the antianginal benefits of bypass surgery versus percutaneous coronary intervention?: implications for future treatment comparisons. Circ Cardiovasc Qual Outcomes. 2012 May;5(3):267-75. doi: 10.1161/CIRCOUTCOMES.111.964585. Epub 2012 Apr 10. PMID 22496114
- [Background] Serruys PW, Farooq V, Vranckx P, Girasis C, Brugaletta S, Garcia-Garcia HM, Holmes DR Jr, Kappetein AP, Mack MJ, Feldman T, Morice MC, Stahle E, James S, Colombo A, Pereda P, Huang J, Morel MA, Van Es GA, Dawkins KD, Mohr FW, Steyerberg EW. A global risk approach to identify patients with left main or 3-vessel disease who could safely and efficaciously be treated with percutaneous coronary intervention: the SYNTAX Trial at 3 years. JACC Cardiovasc Interv. 2012 Jun;5(6):606-17. doi: 10.1016/j.jcin.2012.03.016. PMID 22721655
- [Background] Head SJ, Holmes DR Jr, Mack MJ, Serruys PW, Mohr FW, Morice MC, Colombo A, Kappetein AP; SYNTAX Investigators. Risk profile and 3-year outcomes from the SYNTAX percutaneous coronary intervention and coronary artery bypass grafting nested registries. JACC Cardiovasc Interv. 2012 Jun;5(6):618-25. doi: 10.1016/j.jcin.2012.02.013. PMID 22721656
- [Background] Farooq V, Vergouwe Y, Raber L, Vranckx P, Garcia-Garcia H, Diletti R, Kappetein AP, Morel MA, de Vries T, Swart M, Valgimigli M, Dawkins KD, Windecker S, Steyerberg EW, Serruys PW. Combined anatomical and clinical factors for the long-term risk stratification of patients undergoing percutaneous coronary intervention: the Logistic Clinical SYNTAX score. Eur Heart J. 2012 Dec;33(24):3098-104. doi: 10.1093/eurheartj/ehs295. Epub 2012 Oct 9. PMID 23048195
- [Background] Farooq V, Serruys PW, Bourantas C, Vranckx P, Diletti R, Garcia Garcia HM, Holmes DR, Kappetein AP, Mack M, Feldman T, Morice MC, Colombo A, Morel MA, de Vries T, van Es GA, Steyerberg EW, Dawkins KD, Mohr FW, James S, Stahle E. Incidence and multivariable correlates of long-term mortality in patients treated with surgical or percutaneous revascularization in the synergy between percutaneous coronary intervention with taxus and cardiac surgery (SYNTAX) trial. Eur Heart J. 2012 Dec;33(24):3105-13. doi: 10.1093/eurheartj/ehs367. Epub 2012 Oct 26. PMID 23103663
- [Background] Farooq V, Serruys PW, Garcia-Garcia HM, Zhang Y, Bourantas CV, Holmes DR, Mack M, Feldman T, Morice MC, Stahle E, James S, Colombo A, Diletti R, Papafaklis MI, de Vries T, Morel MA, van Es GA, Mohr FW, Dawkins KD, Kappetein AP, Sianos G, Boersma E. The negative impact of incomplete angiographic revascularization on clinical outcomes and its association with total occlusions: the SYNTAX (Synergy Between Percutaneous Coronary Intervention with Taxus and Cardiac Surgery) trial. J Am Coll Cardiol. 2013 Jan 22;61(3):282-94. doi: 10.1016/j.jacc.2012.10.017. Epub 2012 Dec 19. PMID 23265332
- [Background] Kappetein AP, Head SJ, Morice MC, Banning AP, Serruys PW, Mohr FW, Dawkins KD, Mack MJ; SYNTAX Investigators. Treatment of complex coronary artery disease in patients with diabetes: 5-year results comparing outcomes of bypass surgery and percutaneous coronary intervention in the SYNTAX trial. Eur J Cardiothorac Surg. 2013 May;43(5):1006-13. doi: 10.1093/ejcts/ezt017. Epub 2013 Feb 14. PMID 23413014
- [Background] Mohr FW, Morice MC, Kappetein AP, Feldman TE, Stahle E, Colombo A, Mack MJ, Holmes DR Jr, Morel MA, Van Dyck N, Houle VM, Dawkins KD, Serruys PW. Coronary artery bypass graft surgery versus percutaneous coronary intervention in patients with three-vessel disease and left main coronary disease: 5-year follow-up of the randomised, clinical SYNTAX trial. Lancet. 2013 Feb 23;381(9867):629-38. doi: 10.1016/S0140-6736(13)60141-5. PMID 23439102
- [Background] Farooq V, van Klaveren D, Steyerberg EW, Meliga E, Vergouwe Y, Chieffo A, Kappetein AP, Colombo A, Holmes DR Jr, Mack M, Feldman T, Morice MC, Stahle E, Onuma Y, Morel MA, Garcia-Garcia HM, van Es GA, Dawkins KD, Mohr FW, Serruys PW. Anatomical and clinical characteristics to guide decision making between coronary artery bypass surgery and percutaneous coronary intervention for individual patients: development and validation of SYNTAX score II. Lancet. 2013 Feb 23;381(9867):639-50. doi: 10.1016/S0140-6736(13)60108-7. PMID 23439103
- [Background] Mack MJ, Head SJ, Holmes DR Jr, Stahle E, Feldman TE, Colombo A, Morice MC, Unger F, Erglis A, Stoler R, Dawkins KD, Serruys PW, Mohr FW, Kappetein AP. Analysis of stroke occurring in the SYNTAX trial comparing coronary artery bypass surgery and percutaneous coronary intervention in the treatment of complex coronary artery disease. JACC Cardiovasc Interv. 2013 Apr;6(4):344-54. doi: 10.1016/j.jcin.2012.11.010. Epub 2013 Mar 20. PMID 23523456
- [Background] Farooq V, Girasis C, Magro M, Onuma Y, Morel MA, Heo JH, Garcia-Garcia H, Kappetein AP, van den Brand M, Holmes DR, Mack M, Feldman T, Colombo A, Stahle E, James S, Carrie D, Fournial G, van Es GA, Dawkins KD, Mohr FW, Morice MC, Serruys PW. The CABG SYNTAX Score - an angiographic tool to grade the complexity of coronary disease following coronary artery bypass graft surgery: from the SYNTAX Left Main Angiographic (SYNTAX-LE MANS) substudy. EuroIntervention. 2013 Mar;8(11):1277-85. doi: 10.4244/EIJV8I11A196. PMID 23537954
- [Background] Farooq V, Girasis C, Magro M, Onuma Y, Morel MA, Heo JH, Garcia-Garcia HM, Kappetein AP, van den Brand M, Holmes DR, Mack M, Feldman T, Colombo A, Stahle E, James S, Carrie D, Fournial G, van Es GA, Dawkins KD, Mohr FW, Morice MC, Serruys PW. The coronary artery bypass graft SYNTAX Score: final five-year outcomes from the SYNTAX-LE MANS left main angiographic substudy. EuroIntervention. 2013 Dec;9(8):1009-10. doi: 10.4244/EIJV9I8A170. No abstract available. PMID 23628520
- [Background] Farooq V, Serruys PW, Bourantas CV, Zhang Y, Muramatsu T, Feldman T, Holmes DR, Mack M, Morice MC, Stahle E, Colombo A, de Vries T, Morel MA, Dawkins KD, Kappetein AP, Mohr FW. Quantification of incomplete revascularization and its association with five-year mortality in the synergy between percutaneous coronary intervention with taxus and cardiac surgery (SYNTAX) trial validation of the residual SYNTAX score. Circulation. 2013 Jul 9;128(2):141-51. doi: 10.1161/CIRCULATIONAHA.113.001803. Epub 2013 Jun 13. PMID 23766350
- [Background] Farooq V, Serruys PW, Vranckx P, Bourantas CV, Girasis C, Holmes DR, Kappetein AP, Mack M, Feldman T, Morice MC, Colombo A, Morel MA, de Vries T, Dawkins KD, Mohr FW, James S, Stahle E. Incidence, correlates, and significance of abnormal cardiac enzyme rises in patients treated with surgical or percutaneous based revascularisation: a substudy from the Synergy between Percutaneous Coronary Interventions with Taxus and Cardiac Surgery (SYNTAX) Trial. Int J Cardiol. 2013 Oct 15;168(6):5287-92. doi: 10.1016/j.ijcard.2013.08.013. Epub 2013 Aug 14. PMID 23993326
- [Background] Farooq V, Serruys PW, Zhang Y, Mack M, Stahle E, Holmes DR, Feldman T, Morice MC, Colombo A, Bourantas CV, de Vries T, Morel MA, Dawkins KD, Kappetein AP, Mohr FW. Short-term and long-term clinical impact of stent thrombosis and graft occlusion in the SYNTAX trial at 5 years: Synergy Between Percutaneous Coronary Intervention with Taxus and Cardiac Surgery trial. J Am Coll Cardiol. 2013 Dec 24;62(25):2360-2369. doi: 10.1016/j.jacc.2013.07.106. Epub 2013 Oct 16. PMID 24140677
- [Background] Girasis C, Farooq V, Diletti R, Muramatsu T, Bourantas CV, Onuma Y, Holmes DR, Feldman TE, Morel MA, van Es GA, Dawkins KD, Morice MC, Serruys PW. Impact of 3-dimensional bifurcation angle on 5-year outcome of patients after percutaneous coronary intervention for left main coronary artery disease: a substudy of the SYNTAX trial (synergy between percutaneous coronary intervention with taxus and cardiac surgery). JACC Cardiovasc Interv. 2013 Dec;6(12):1250-60. doi: 10.1016/j.jcin.2013.08.009. PMID 24355115
- [Background] Morice MC, Serruys PW, Kappetein AP, Feldman TE, Stahle E, Colombo A, Mack MJ, Holmes DR, Choi JW, Ruzyllo W, Religa G, Huang J, Roy K, Dawkins KD, Mohr F. Five-year outcomes in patients with left main disease treated with either percutaneous coronary intervention or coronary artery bypass grafting in the synergy between percutaneous coronary intervention with taxus and cardiac surgery trial. Circulation. 2014 Jun 10;129(23):2388-94. doi: 10.1161/CIRCULATIONAHA.113.006689. Epub 2014 Apr 3. PMID 24700706
- [Background] Head SJ, Davierwala PM, Serruys PW, Redwood SR, Colombo A, Mack MJ, Morice MC, Holmes DR Jr, Feldman TE, Stahle E, Underwood P, Dawkins KD, Kappetein AP, Mohr FW. Coronary artery bypass grafting vs. percutaneous coronary intervention for patients with three-vessel disease: final five-year follow-up of the SYNTAX trial. Eur Heart J. 2014 Oct 21;35(40):2821-30. doi: 10.1093/eurheartj/ehu213. Epub 2014 May 21. PMID 24849105
- [Derived] Serruys PW, Ninomiya K, Revaiah PC, Gao C, Garg S, van Klaveren D, Onuma Y, Kappetein AP, Davierwala P, Mack M, Thuijs DJFM, Taggart DP, Milojevic M. Ten-year survival benefit and appropriateness of surgical versus percutaneous revascularization in synergy between percutaneous coronary intervention with Taxus and cardiac surgery randomized trial. Eur J Cardiothorac Surg. 2024 Nov 4;66(5):ezae391. doi: 10.1093/ejcts/ezae391. PMID 39447048
- [Derived] Ninomiya K, Serruys PW, Garg S, Kageyama S, Kotoku N, Masuda S, Revaiah PC, O'leary N, Kappetein AP, Mack MJ, Holmes DR, Davierwala PM, Mohr FW, Thuijs DJFM, Onuma Y; SYNTAX Extended Survival (SYNTAXES) Investigators. gamma-Glutamyl Transferase and Long-Term Survival in the SYNTAXES Trial: Is It Just the Liver? J Am Heart Assoc. 2024 Apr 16;13(8):e032276. doi: 10.1161/JAHA.123.032276. Epub 2024 Apr 2. PMID 38563386
- [Derived] Ninomiya K, Kageyama S, Garg S, Masuda S, Kotoku N, Revaiah PC, O'leary N, Onuma Y, Serruys PW; SYNTAX Extended Survival Investigators. Can machine learning unravel unsuspected, clinically important factors predictive of long-term mortality in complex coronary artery disease? A call for 'big data'. Eur Heart J Digit Health. 2023 Feb 28;4(3):275-278. doi: 10.1093/ehjdh/ztad014. eCollection 2023 May. PMID 37265868
- [Derived] Wang R, Lunardi M, Hara H, Gao C, Ono M, Davierwala PM, Holmes DR, Mohr FW, Curzen N, Burzotta F, van Geuns RJ, Kappetein AP, Head SJ, Thuijs DJFM, Tao L, Garg S, Onuma Y, Wijns W, Serruys PW. Impact of repeat revascularization within 5 years on 10-year mortality after percutaneous or surgical revascularization. Clin Res Cardiol. 2023 Sep;112(9):1302-1311. doi: 10.1007/s00392-023-02211-6. Epub 2023 May 8. PMID 37150783
- [Derived] Ono M, Serruys PW, Kawashima H, Lunardi M, Wang R, Hara H, Gao C, Garg S, O'Leary N, Wykrzykowska JJ, Piek JJ, Holmes DR, Morice MC, Kappetein AP, Noack T, Davierwala PM, Spertus JA, Cohen DJ, Onuma Y; SYNTAX Extended Survival Investigators. Impact of residual angina on long-term clinical outcomes after percutaneous coronary intervention or coronary artery bypass graft for complex coronary artery disease. Eur Heart J Qual Care Clin Outcomes. 2023 Aug 7;9(5):490-501. doi: 10.1093/ehjqcco/qcac052. PMID 36001991
- [Derived] Ono M, Serruys PW, Garg S, Kawashima H, Gao C, Hara H, Lunardi M, Wang R, O'Leary N, Wykrzykowska JJ, Piek JJ, Mack MJ, Holmes DR, Morice MC, Kappetein AP, Thuijs DJFM, Noack T, Mohr FW, Davierwala PM, Spertus JA, Cohen DJ, Onuma Y; SYNTAX Extended Survival Investigators. Effect of Patient-Reported Preprocedural Physical and Mental Health on 10-Year Mortality After Percutaneous or Surgical Coronary Revascularization. Circulation. 2022 Oct 25;146(17):1268-1280. doi: 10.1161/CIRCULATIONAHA.121.057021. Epub 2022 Jul 18. PMID 35862109
- [Derived] Ono M, Hara H, Gao C, Kawashima H, Wang R, O'Leary N, Wykrzykowska JJ, Piek JJ, Mack MJ, Holmes D, Morice MC, Head S, Kappetein AP, Noack T, Davierwala PM, Mohr FW, Garg S, Onuma Y, Serruys PW; SYNTAX Extended Survival Investigators. Mortality after multivessel revascularisation involving the proximal left anterior descending artery. Heart. 2022 Oct 28;108(22):1784-1791. doi: 10.1136/heartjnl-2022-320934. PMID 35732441
- [Derived] Kawashima H, Serruys PW, Hara H, Ono M, Gao C, Wang R, Garg S, Sharif F, de Winter RJ, Mack MJ, Holmes DR, Morice MC, Kappetein AP, Thuijs DJFM, Milojevic M, Noack T, Mohr FW, Davierwala PM, Onuma Y; SYNTAX Extended Survival Investigators. 10-Year All-Cause Mortality Following Percutaneous or Surgical Revascularization in Patients With Heavy Calcification. JACC Cardiovasc Interv. 2022 Jan 24;15(2):193-204. doi: 10.1016/j.jcin.2021.10.026. Epub 2021 Dec 29. PMID 34973904
- [Derived] Hara H, Kawashima H, Ono M, Takahashi K, Mack MJ, Holmes DR Jr, Morice MC, Davierwala PM, Mohr FW, Thuijs DJFM, Kappetein AP, O'Leary N, van Klaveren D, Onuma Y, Serruys PW. Impact of preprocedural biological markers on 10-year mortality in the SYNTAXES trial. EuroIntervention. 2022 Apr 22;17(18):1477-1487. doi: 10.4244/EIJ-D-21-00415. PMID 34669586
- [Derived] Thuijs DJFM, Davierwala P, Milojevic M, Deo SV, Noack T, Kappetein AP, Serruys PW, Mohr FW, Morice MC, Mack MJ, Stahle LEGE, Verberkmoes NJ, Holmes DR, Head SJ; SYNTAX Extended Survival Investigators. Long-term survival after coronary bypass surgery with multiple versus single arterial grafts. Eur J Cardiothorac Surg. 2022 Mar 24;61(4):925-933. doi: 10.1093/ejcts/ezab392. PMID 34618017
- [Derived] Wang R, Garg S, Gao C, Kawashima H, Ono M, Hara H, van Geuns RJ, Morice MC, Davierwala PM, Kappetein AP, Holmes DR, Wijns W, Tao L, Onuma Y, Serruys PW. Impact of established cardiovascular disease on 10-year death after coronary revascularization for complex coronary artery disease. Clin Res Cardiol. 2021 Oct;110(10):1680-1691. doi: 10.1007/s00392-021-01922-y. Epub 2021 Aug 25. PMID 34432113
- [Derived] Davierwala PM, Gao C, Thuijs DJFM, Wang R, Hara H, Ono M, Noack T, Garg S, O'leary N, Milojevic M, Kappetein AP, Morice MC, Mack MJ, van Geuns RJ, Holmes DR, Gaudino M, Taggart DP, Onuma Y, Mohr FW, Serruys PW; SYNTAX Extended Survival Investigators. Single or multiple arterial bypass graft surgery vs. percutaneous coronary intervention in patients with three-vessel or left main coronary artery disease. Eur Heart J. 2022 Mar 31;43(13):1334-1344. doi: 10.1093/eurheartj/ehab537. PMID 34405875
- [Derived] Wang R, Serruys PW, Gao C, Hara H, Takahashi K, Ono M, Kawashima H, O'leary N, Holmes DR, Witkowski A, Curzen N, Burzotta F, James S, van Geuns RJ, Kappetein AP, Morel MA, Head SJ, Thuijs DJFM, Davierwala PM, O'Brien T, Fuster V, Garg S, Onuma Y. Ten-year all-cause death after percutaneous or surgical revascularization in diabetic patients with complex coronary artery disease. Eur Heart J. 2021 Dec 28;43(1):56-67. doi: 10.1093/eurheartj/ehab441. PMID 34405232
- [Derived] Ono M, Kawashima H, Hara H, Mancone M, Mack MJ, Holmes DR, Morice MC, Kappetein AP, Thuijs DJFM, Noack T, Mohr FW, Davierwala PM, Onuma Y, Serruys PW; SYNTAX Extended Survival Investigators. Impact of major infections on 10-year mortality after revascularization in patients with complex coronary artery disease. Int J Cardiol. 2021 Oct 15;341:9-12. doi: 10.1016/j.ijcard.2021.08.013. Epub 2021 Aug 8. PMID 34375706
- [Derived] Kawashima H, Serruys PW, Ono M, Hara H, O'Leary N, Mack MJ, Holmes DR, Morice MC, Head SJ, Kappetein AP, Thuijs DJFM, Milojevic M, Noack T, Mohr FW, Davierwala PM, Sharif F, McEvoy JW, Onuma Y; SYNTAX Extended Survival Investigators. Impact of Optimal Medical Therapy on 10-Year Mortality After Coronary Revascularization. J Am Coll Cardiol. 2021 Jul 6;78(1):27-38. doi: 10.1016/j.jacc.2021.04.087. PMID 34210411
- [Derived] Ono M, Serruys PW, Hara H, Kawashima H, Gao C, Wang R, Takahashi K, O'Leary N, Wykrzykowska JJ, Sharif F, Piek JJ, Garg S, Mack MJ, Holmes DR, Morice MC, Head SJ, Kappetein AP, Thuijs DJFM, Noack T, Davierwala PM, Mohr FW, Cohen DJ, Onuma Y; SYNTAX Extended Survival Investigators. 10-Year Follow-Up After Revascularization in Elderly Patients With Complex Coronary Artery Disease. J Am Coll Cardiol. 2021 Jun 8;77(22):2761-2773. doi: 10.1016/j.jacc.2021.04.016. PMID 34082905
- [Derived] Takahashi K, Serruys PW, Gao C, Ono M, Wang R, Thuijs DJFM, Mack MJ, Curzen N, Mohr FW, Davierwala P, Milojevic M, Wykrzykowska JJ, de Winter RJ, Sharif F, Onuma Y, Head SJ, Kappetein AP, Morice MC, Holmes DR Jr; SYNTAX Extended Survival Study Investigators. Ten-Year All-Cause Death According to Completeness of Revascularization in Patients With Three-Vessel Disease or Left Main Coronary Artery Disease: Insights From the SYNTAX Extended Survival Study. Circulation. 2021 Jul 13;144(2):96-109. doi: 10.1161/CIRCULATIONAHA.120.046289. Epub 2021 May 20. PMID 34011163
- [Derived] Wang R, Tomaniak M, Takahashi K, Gao C, Kawashima H, Hara H, Ono M, van Klaveren D, van Geuns RJ, Morice MC, Davierwala PM, Mack MJ, Witkowski A, Curzen N, Berti S, Burzotta F, James S, Kappetein AP, Head SJ, Thuijs DJFM, Mohr FW, Holmes DR, Tao L, Onuma Y, Serruys PW. Impact of chronic obstructive pulmonary disease on 10-year mortality after percutaneous coronary intervention and bypass surgery for complex coronary artery disease: insights from the SYNTAX Extended Survival study. Clin Res Cardiol. 2021 Jul;110(7):1083-1095. doi: 10.1007/s00392-021-01833-y. Epub 2021 Mar 12. PMID 33710385
- [Derived] Takahashi K, Thuijs DJFM, Gao C, Ono M, Holmes DR, Mack MJ, Morice MC, Mohr FW, Curzen N, Davierwala PM, Milojevic M, Dawkins KD, Wykrzykowska JJ, de Winter RJ, McEvoy JW, Onuma Y, Head SJ, Kappetein AP, Serruys PW; SYNTAX Extended Survival Study Investigators. Ten-year all-cause mortality according to smoking status in patients with severe coronary artery disease undergoing surgical or percutaneous revascularization. Eur J Prev Cardiol. 2022 Mar 11;29(2):312-320. doi: 10.1093/eurjpc/zwaa089. PMID 33624046
- [Derived] Kawashima H, Takahashi K, Ono M, Hara H, Wang R, Gao C, Sharif F, Mack MJ, Holmes DR, Morice MC, Head SJ, Kappetein AP, Thuijs DJFM, Milojevic M, Noack T, Mohr FW, Davierwala PM, Serruys PW, Onuma Y; SYNTAX Extended Survival Investigators. Mortality 10 Years After Percutaneous or Surgical Revascularization in Patients With Total Coronary Artery Occlusions. J Am Coll Cardiol. 2021 Feb 9;77(5):529-540. doi: 10.1016/j.jacc.2020.11.055. PMID 33538250
- [Derived] Wang R, Takahashi K, Garg S, Thuijs DJFM, Kappetein AP, Mack MJ, Morice MC, Mohr FW, Curzen N, Davierwala P, Milojevic M, van Geuns RJ, Head SJ, Onuma Y, Holmes DR Jr, Serruys PW. Ten-year all-cause death following percutaneous or surgical revascularization in patients with prior cerebrovascular disease: insights from the SYNTAX Extended Survival study. Clin Res Cardiol. 2021 Oct;110(10):1543-1553. doi: 10.1007/s00392-020-01802-x. Epub 2021 Jan 30. PMID 33517534
- [Derived] Hara H, Serruys PW, Takahashi K, Kawashima H, Ono M, Gao C, Wang R, Mohr FW, Holmes DR, Davierwala PM, Head SJ, Thuijs DJFM, Milojevic M, Kappetein AP, Garg S, Onuma Y, Mack MJ; SYNTAX Extended Survival Investigators. Impact of Peri-Procedural Myocardial Infarction on Outcomes After Revascularization. J Am Coll Cardiol. 2020 Oct 6;76(14):1622-1639. doi: 10.1016/j.jacc.2020.08.009. PMID 33004127
- [Derived] Hara H, Takahashi K, van Klaveren D, Wang R, Garg S, Ono M, Kawashima H, Gao C, Mack M, Holmes DR, Morice MC, Head SJ, Kappetein AP, Thuijs DJFM, Onuma Y, Noack T, Mohr FW, Davierwala PM, Serruys PW; SYNTAX Extended Survival Investigators. Sex Differences in All-Cause Mortality in the Decade Following Complex Coronary Revascularization. J Am Coll Cardiol. 2020 Aug 25;76(8):889-899. doi: 10.1016/j.jacc.2020.06.066. PMID 32819461
- [Derived] Thuijs DJFM, Kappetein AP, Serruys PW, Mohr FW, Morice MC, Mack MJ, Holmes DR Jr, Curzen N, Davierwala P, Noack T, Milojevic M, Dawkins KD, da Costa BR, Juni P, Head SJ; SYNTAX Extended Survival Investigators. Percutaneous coronary intervention versus coronary artery bypass grafting in patients with three-vessel or left main coronary artery disease: 10-year follow-up of the multicentre randomised controlled SYNTAX trial. Lancet. 2019 Oct 12;394(10206):1325-1334. doi: 10.1016/S0140-6736(19)31997-X. Epub 2019 Sep 2. PMID 31488373